CLINICAL TRIAL: NCT01162317
Title: Novel Approaches to Sleep Difficulties: Application in Mild TBI
Brief Title: AcuSleep in Mild Traumatic Brain Injury (TBI)
Acronym: AcuTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: B6924-W
Record Dates: First submitted 2010-06-15; First posted 2010-07-14 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Brain Injuries, Traumatic; Sleeplessness
Keywords: Acupuncture; Sleep; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Sleep Initiation and Maintenance Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: sham acupuncture (Active Comparator): sham acupuncture
  Interventions: Other: Sham Acupuncture
- Arm 2: acupuncture (Experimental): acupuncture
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Treatments will be performed by the PI, who is a licensed physician acupuncturist and has practiced acupuncture independently for 5 years with about 4000 patient/visit treatment history. A total of 10 acupuncture treatments represents a reasonable approach to optimal duration of treatment. Acupoint selection will be based on a combination of standardization and individualization for best treatment effects. At least 5 standardized body and auricular acupoints will be selected. Standardized sterile, disposable acupuncture needles will be applied for 20 minutes.
  Arms: Arm 2: acupuncture
Other: Sham Acupuncture — Treatments will be performed by the PI, who is a licensed physician acupuncturist and has practiced acupuncture independently for 5 years with about 4000 patient/visit treatment history. A total of 10 acupuncture treatments represent a reasonable approach to optimal duration of treatment. Acupoint selection will be based on a combination of standardization and individualization for best treatment effects. At least 5 standardized body and auricular acupoints will be selected. Standardized sterile, disposable acupuncture needles will be applied for 20 minutes. Each sham or real acupuncture needle will be applied through a tube as sham needles have blunt tip and telescopic shaft, the visual effect and percutaneous sensation of sham needle mimic the real needle penetration.
  Arms: Arm 1: sham acupuncture

SUMMARY:
Objective: To evaluate real acupuncture, as compare to sham acupuncture, in improving persistent sleep difficulties in veterans with mild traumatic brain injury (mTBI) Design: Randomized, blinded, sham-controlled clinical trial Setting: Outpatient clinic at a major VA medical center in Southeast USA Participants: Sixty veterans aged 24-55 (mean 40) with history of mTBI at least 3-month and beyond, suffering from sleep difficulties refractory to regular care and sleep education, as indicated by a global Pittsburgh Sleep Quality Index (PSQI) score of 14.25 + 3.23 pre-intervention (baseline). They were randomized into 2 groups, real acupuncture versus sham acupuncture, and stratified by Post-traumatic stress disorder (PTSD) diagnosed by PTSD CheckList - Military Version (PCL-M).

Intervention: Real or sham acupuncture with both standardized and individualized acupoints selection. All subjects were informed that the treatments, if effective, may improve symptoms such as pain, anxiety or depression other than sleep; real acupuncture may not be effective in some individuals, and sham acupuncture may as well be effective by mind-body interactions.

Outcome Measures: Primary outcome measure was global PSQI score change after intervention as compared to baseline. Secondary outcome measure was wrist-actigraphy sleep latency, sleep efficiency, wake after sleep onset (WASO), and sleep duration. PTSD was analyzed as a co-variant.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 55; and,
* Meeting the diagnosis criteria for mild traumatic brain injury as listed above at the time of injury; and,
* At or over 3 months post injury; and,
* With untreated sleep complaints (Pittsburgh Sleep Quality Index [PSQI] > 8, sleep difficulties at least 4x per week in the past month, average sleep duration of 6 hours or less); and,
* Has the capacity to give informed consent.
* Agree to attend 13 clinic visits

Exclusion Criteria:

* Same sleep complaints present prior to traumatic brain injury; or,
* Diagnosis of obstructive sleep apnea (OSA) by prior sleep study; or,
* With a non-daytime work-schedule; or,
* With prior acupuncture experience for the treatment of sleep difficulties or with acupuncture treatment within 3 months; or,
* History of bleeding diathesis or currently on anticoagulation with international normalized ratio (INR) over 2.5; or,
* Severe depression with Beck Depression Score of 29 and above; or,
* Moderate and severe alcohol users.
* Does not have a permanent address

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07-05 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2017-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Huang, MD PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang W, Johnson TM, Kutner NG, Halpin SN, Weiss P, Griffiths PC, Bliwise DL. Acupuncture for Treatment of Persistent Disturbed Sleep: A Randomized Clinical Trial in Veterans With Mild Traumatic Brain Injury and Posttraumatic Stress Disorder. J Clin Psychiatry. 2018 Dec 11;80(1):18m12235. doi: 10.4088/JCP.18m12235. PMID 30549498

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Sham Acupuncture | Arm 2: Acupuncture
Started | 30 | 30
Completed | 27 | 28
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Sham Acupuncture | Arm 2: Acupuncture | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (10.3) | 39.6 (9.7) | 39.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 22 | 24 | 46
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
Pittsburgh Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: units on a scale] — In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. Only global PSQI scores were used for this study.
  units on a scale | 14.33 (3.10) | 14.17 (3.41) | 14.26 (3.20)

OUTCOME MEASURES:

1. Primary Outcome: PSQI Change
Description: change of global PSQI score as compared to baseline The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval.
  The PSQI global score has a possible range of 0-21 points. Any score above 5 is considered insomnia. The higher the score the worse the condition.
Time Frame: Baseline and post-intervention
Measure: Mean (Standard Deviation); unit: change of points from baseline
Arm/Group | Arm 1: Sham Acupuncture | Arm 2: Acupuncture
Number analyzed (Participants) | 30 | 30
change of points from baseline | -2.38 (3.41) | -4.43 (3.86)

2. Secondary Outcome: Wrist Actigraphy (an Objective Sleep Measure) Sleep Efficiency
Description: Wrist actigraphy is a non-invasive method of continuously monitoring gross body activities when a watch-like actimetry sensor is worn at the non-dominant wrist. An algorithm has been developed to assess sleep/wake behavior. Specifically in this study, we used Respironics® actiwatches for data collection. Subjects were asked to wear the actiwatches for a consecutive week at baseline and then at post-intervention, and the actiwatches were taken off only during showers. Wrist actigraphy was examined in association with sleep diary the subjects were to keep for the weeks of monitoring. Threshold-based method algorithm for data interpretation was provided by Respironics® Actiware Software. Medium level threshold was set to detect Wake and Sleep; sleep interval detection algorithm was set for 3 minutes of immobile minutes for Sleep Onset and 5 minutes of immobile minutes for Sleep End. Sleep efficiency is sleep duration divided by total bed time (both in minutes), times 100%.
Time Frame: pre-intervention, post-intervention (1wk of recording each)
Population: All obtained actigraphy data were analyzed. This form doesn't allow specific indication of sample sizes. Therefore, here overall numbers of participants analyzed were the same as the maximal potential.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Arm 1: Sham Acupuncture | Arm 2: Acupuncture
Number analyzed (Participants) | 30 | 30
percentage
  Pre-intervention: number analyzed (Participants) | 30 | 20
  Pre-intervention | 73.57 (13.21) | 72.57 (16.41)
  Post-intervention: number analyzed (Participants) | 19 | 30
  Post-intervention | 67.94 (13.28) | 76.68 (12.18)

ADVERSE EVENTS:
Arm/Group | Arm 1: Sham Acupuncture | Arm 2: Acupuncture
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 8/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Sham Acupuncture (N=30) | Arm 2: Acupuncture (N=30)
Needle site pain (Skin and subcutaneous tissue disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes